CLINICAL TRIAL: NCT00671398
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Multicenter, Single-Dose Study of TAK-375 in Healthy Adult Volunteers in a Sleep Lab Model of Transient Insomnia
Brief Title: Efficacy of Ramelteon on Transient Insomnia in Healthy Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-02-TL-375-023; U1111-1114-8626 (Registry Identifier: WHO)
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Transient Insomnia
Keywords: Insomnia; Sleep Disorder; Drug Therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ramelteon 8 mg QD (Experimental)
  Interventions: Drug: Ramelteon
- Ramelteon 16 mg QD (Experimental)
  Interventions: Drug: Ramelteon
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon — Ramelteon 8 mg, tablets, orally for one night only.
  Other Names: Rozerem™; TAK-375
  Arms: Ramelteon 8 mg QD
Drug: Ramelteon — Ramelteon 16 mg, tablets, orally for one night only
  Other Names: Rozerem™; TAK-375
  Arms: Ramelteon 16 mg QD
Drug: Placebo — Ramelteon placebo-matching tablets, orally for one night only
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Ramelteon, once daily (QD), in healthy subjects within a sleep lab.

DETAILED DESCRIPTION:
Insomnia is characterized by difficulties initiating and maintaining sleep, or of non-restorative and non-refreshing sleep. Transient insomnia affects approximately one-third to one-half of the US population, based on the results of 2 surveys of representative samples of the adult US population conducted by the Gallup Organization in which respondents were asked if they had "ever had difficulty sleeping." Based on reports of "regular" or "frequent" sleep difficulty, results from the same studies suggest that approximately one-tenth of the US population experiences chronic insomnia. The ideal treatment for insomnia would reduce the latency to onset of sleep and increase total sleep time, without a negative impact on sleep architecture and without safety concerns or next-day effects.

Ramelteon is a selective melatonin-1 receptor agonist under global development by Takeda Chemical Industries, Ltd., for the treatment of transient and chronic insomnia and for the treatment of Circadian Rhythm Sleep Disorders.

This study is being conducted to evaluate the safety and efficacy of a single dose of Ramelteon in normal healthy subjects in a sleep lab model of transient insomnia. Participation is this study is anticipated to be about 3 weeks.

ELIGIBILITY:
Inclusion Criteria

* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Habitual bedtime is between 8:30 p.m. and 12:00 a.m.
* Sleeps 6.5 to 8 hours per night and has a subjective sleep latency of less than or equal to 30 minutes.
* Body mass index between 18 and 34, inclusive.

Exclusion Criteria:

* Any history of insomnia.
* Spent one or more nights in a sleep laboratory.
* Epworth Sleepiness Scale score of greater than 10.
* Known hypersensitivity to Ramelteon or related compounds, including melatonin.
* Previously participated in a study involving Ramelteon.
* Participated in any other investigational study and/or taken any investigational drug within 30 days or five half-lives prior to Day 1, whichever is longer.
* Sleep schedule changes required by employment (ie, shift work) within three months preceding Day 1 or has flown across greater than three time zones within seven days prior to screening.
* Participated in a weight loss program or substantially altered their exercise routine within 30 days prior to Day 1.
* History of seizures, sleep apnea, chronic obstructive pulmonary disease, restless leg syndrome, schizophrenia, bipolar disorder, mental retardation, or cognitive disorder.
* History of a psychiatric disorder (including anxiety or depression) within the past 12 months.
* History of drug addiction or drug abuse within the past 12 months.
* Any physical or psychiatric disorder that may be associated with sleep disturbance.
* History of alcohol abuse within the past 12 months, as defined in Diagnostic and Statistical Manual of Mental Disorders, 4th Edition Revised and/or regularly consumes 4 or more alcoholic drinks per day.
* Current significant neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, hematologic or metabolic disease.
* Uses tobacco products during nightly awakenings.
* Any clinically important abnormal finding as determined by a medical history, physical examination, electrocardiogram, or clinical laboratory tests, as determined by the investigator.
* Positive hepatitis panel.
* Positive urine drug screen including alcohol at screening or a positive breathalyzer test at check-in.
* Any additional condition(s) that in the investigator's opinion would

  * affect sleep-wake function
  * prohibit the subject from completing the study
  * not be in the best interest of the subject.
* Is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication, including:

  * Anxiolytics
  * Hypnotics
  * Antidepressants
  * Anticonvulsants
  * Sedating H1 antihistamines
  * Systemic steroids
  * Respiratory stimulants (eg, theophylline)
  * Decongestants
  * Over-the-counter and prescription stimulants
  * Over-the-counter and prescription diet aids
  * Central nervous system active drugs
  * Narcotic analgesics
  * All beta blockers
  * St. John's Wort
  * Kava-kava
  * gingko biloba

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 289 (Actual)
Dates: Start 2002-12; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Latency to Persistent Sleep from 1 night of polysomnography (PSG) recording in a sleep laboratory. | Day 1

SECONDARY OUTCOMES:
Total Sleep Time. | Days 1 and 2.
Sleep Efficiency. | Days 1 and 2.
Wake Time after Persistent Sleep Onset. | Days 1 and 2.
Number of Awakenings after Persistent Sleep. | Days 1 and 2.
Subjective Sleep Latency. | Day 2
Subjective Total Sleep Time. | Day 2
Subjective Sleep Quality. | Day 2
Subjective Wake Time after Sleep Onset. | Day 2
Subjective Number of Awakenings. | Day 2
Subjective Ease of Falling Back to Sleep after Awakening. | Day 2
Stage 1 Nonrapid Eye Movement (NREM) Sleep | Day 2.
Stage 2 Nonrapid Eye Movement (NREM) Sleep | Day 2.
Stage 3/4 Nonrapid Eye Movement (NREM) Sleep | Day 2.
Latency to Rapid Eye Movement (REM) Sleep | Day 2.
Percentage of Total Sleep Time in REM Sleep | Day 2.

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science, Study Director — Takeda
Locations (12):
- United States (12):
  - Palm Springs, California
  - San Diego, California
  - Miami, Florida
  - Pembroke Pines, Florida
  - Atlanta, Georgia
  - Overland Park, Kansas
  - New York, New York
  - Rochester, New York
  - Cincinnati, Ohio
  - Dublin, Ohio
  - Columbia, South Carolina
  - Houston, Texas

REFERENCES:
- [Result] Zammit G, Schwartz H, Roth T, Wang-Weigand S, Sainati S, Zhang J. The effects of ramelteon in a first-night model of transient insomnia. Sleep Med. 2009 Jan;10(1):55-9. doi: 10.1016/j.sleep.2008.04.010. Epub 2008 Aug 8. PMID 18691937
- See also: Rozerem Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI